CLINICAL TRIAL: NCT00166621
Title: Early Pharmacotherapy Aimed at Neuroplasticity in Autism : Safety and Efficacy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chugani, Diane C. (Individual)
Responsible Party: Diane C Chugani, Wayne State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PPRU 10659s
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Autism
Keywords: Autism; Neuroplasticity
MeSH Terms: conditions — Autistic Disorder | interventions — Buspirone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Buspirone

SUMMARY:
The purpose of this study is to determine the efficacy, safety, and population pharmacokinetics and determinants of drug responses to buspirone in children with autism using a randomized, double blind, cross over study in children ages 2 to 6 years.

DETAILED DESCRIPTION:
Autism is a neurodevelopmental disorder defined as qualitative impairment in social interaction and communication and restrictive stereotype patterns of behavior, interests and activities. Pharmacological agents are being increasingly used off label in very young autistic children, and there is virtually no data regarding the pharmacokinetics, safety or efficacy of these agents in young children.

The approach in this study differs from pharmacotherapy studies of autism carried out thus far in several ways:

* the rationale underlying our approach is based upon an attempt to alter synaptic plasticity during postnatal development, focusing on very young children
* are integrating our drug trial with a PG study evaluating whether buspirone response is related to expression of genes involved in serotoninergic neurotransmission
* will assess these variables together with in vivo assessment of serotonin synthesis capacity with PET.

This is a prospective, randomized, double blind, crossover study where children will be stratified by age into two groups. Treatment will last for 12 weeks with dosing twice a day. Parent ratings, cognitive tests and blood sampling will occur throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Meet study definition for the diagnosis of autistic disorder
* Age 2 to 6 (male or female)
* Informed Consent

Exclusion Criteria:

* Clinical or lab evidence of renal or hepatic disease
* Treatment with any medication known to alter the activity of the CYP3A4 enzyme including ketoconazole, itraconazole, grapefruit juice, erythromycin, clarithromycin, cimetidine, verapamil, diltiazem, rifampin, phenytoin, phenobarbital, or carbamazepine within the previous 3 months
* Use of centrally acting drugs during the 6 weeks prior or during the study
* Presence or history of neurological disorders, including seizure disorders

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20
Dates: Start 2004-03; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Safety will be measured by obtaining clinical laboratory tests, vital signs and evaluating probably or definitely related adverse events.
Population pharmacokinetics will be conducted to measure plasma concentrations in relation to the drug responses to buspirone.
The primary efficacy outcome will be the overall severity score from the Clinical Global Impressions assessment obtained from two raters, (parent and examiner)
Comparisons of allele, and genotype frequencies between responders and non-responders will be done for each polymorphism using Fisher's exact test to best predict response to buspirone.

CONTACTS AND LOCATIONS:
Locations (1):
- PET Center/Children's Hospital of Michigan, Detroit, Michigan, United States